CLINICAL TRIAL: NCT04428645
Title: Assessment of a Decision Support Tool in Participants With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jessica Castle, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19950
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- DailyDose Decision Support (Experimental): Subjects will use DailyDose decision support for 8 weeks at home.
  Interventions: Device: DailyDose Decision Support

INTERVENTIONS:
Device: DailyDose Decision Support — DailyDose provides on-demand, real-time dosing recommendations for insulin meal boluses and basal insulin doses as well as the option to receive recommendations for meals and exercise. DailyDose is an information system comprised of (1) a smart phone app that both collects continuous glucose measurement (CGM) data, insulin data, and fitness data and presents suggestions back to the user, (2) a cloud based information system that stores the raw data and relays suggestions to the user, (3) a glucoregulatory model, automatically personalized for each user, that resides on a cloud server and is fit with the user's individual glucose data, and (4) an adaptive agent that provides insulin dosing options and suggestions as well as meal and exercise recommendations to the user based on the subject's own outcomes and simulations done on the glucoregulatory model.

SUMMARY:
Type 1 diabetes (T1D) is a complex disease with a high risk of both hyper- and hypoglycemia which can lead to severe acute and chronic complications. The burden and complexity of managing T1D results in the majority of people not reaching adequate glycemic control. Our team has developed a smartphone based application, DailyDose, that combines continuous glucose monitoring data and insulin data to provide decision support for subjects with type 1 diabetes taking multiple daily injections (MDI). DailyDose provides on-demand, real-time dosing recommendations for insulin doses prior to meals and to correct hyperglycemia. DailyDose analyzes glucose patterns and provides weekly recommendations to the patient on insulin settings including carbohydrate ratios and correction factors. As needed, DailyDose will make weekly recommendations to change basal insulin. For subject safety, study investigators will set constraints on settings for short and long acting insulin during the onboarding process. DailyDose will not be able to recommend insulin dose changes above or below the set safety thresholds. DailyDose also provides recommendations on carbohydrate intake for exercise and includes hypoglycemia and hyperglycemia alarms.

DETAILED DESCRIPTION:
Subjects will be on study for 10 weeks. Subjects will begin the study with a training visit on the Dexcom G6 CGM system and the InPen and Clipsulin smart insulin pens. Subjects will use these devices for the next 14 days at home. Subjects will return to OHSU at the end of the 14 days for a training on using the DailyDose system. Subjects will then return home to use the DailyDose system for 8 weeks. Sensor glucose, exercise, insulin and meal data will be collected during the DailyDose portion of the study in order to produce recommendations for insulin dosing. Subjects will receive up to 4 recommendations every 7 days. Subjects will also receive recommendations for exercise based on the PEAK exercise guidelines.

Subjects will wear the Dexcom G6 and an Apple Watch physical activity monitor for the entire study. Insulin data will be collected using the InPen for aspart insulin and Clipsulin for the long acting insulin. Subjects will complete a 30 minute aerobic exercise video at home once per week. Subjects will also be asked to complete two additional exercise sessions on their own at home, one aerobic session and the other whatever type of exercise they would normally do (aerobic, resistance etc.). Subjects will use the bolus calculator within the DailyDose app. Subjects will be instructed to test capillary blood glucose (CBG) after exercise, for symptoms of hypoglycemia or hypoglycemia alerts and again 15 minutes after rescue carbohydrate treatment until CBG >70 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus for at least 1 year.
* Male or female subjects 18 to 60 years of age.
* Physically willing and able to perform 30 min of exercise (as determined by the investigator after reviewing the subject's activity level).
* Use of multiple daily insulin injections (MDI) for at least 4 weeks at time of screening visit.
* A1C 7.0-10.0% at the time of screening.
* Willingness to follow all study procedures, including attending all clinic visits.
* Willingness to sign informed consent and HIPAA documents.

Exclusion Criteria:

* Female of childbearing potential who is pregnant or intending to become pregnant or breast-feeding, or is not using adequate contraceptive methods. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
* Any cardiovascular disease, defined as a clinically significant EKG abnormality at the time of screening or any history of: stroke, heart failure, myocardial infarction, angina pectoris, or coronary arterial bypass graft or angioplasty. Diagnosis of 2nd or 3rd degree heart block or any non-physiological arrhythmia judged by the investigator to be exclusionary.
* Renal insufficiency (GFR < 60 ml/min, using the MDRD equation as reported by the OHSU laboratory).
* Liver failure, cirrhosis, or any other liver disease that compromises liver function as determined by the investigator.
* History of severe hypoglycemia during the past 6 months prior to screening visit or hypoglycemia unawareness as judged by the investigator. Subjects will complete a hypoglycemia awareness questionnaire. Subjects will be excluded for four or more R responses.
* Any active infection.
* Known or suspected abuse of alcohol, narcotics, or illicit drugs.
* Seizure disorder.
* Active foot ulceration.
* Peripheral arterial disease.
* Major surgical operation within 30 days prior to screening.
* Use of an investigational drug within 30 days prior to screening.
* Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
* Allergy to aspart insulin.
* Current administration of oral or parenteral corticosteroids.
* Any life threatening disease, including malignant neoplasms and medical history of malignant neoplasms within the past 5 years prior to screening (except basal and squamous cell skin cancer).
* Current use of any medication intended to lower glucose other than insulin (ex. use of liraglutide).
* Vision impairment which in the opinion of the investigator would preclude the use of the smart phone application.
* A positive response to any of the questions from the Physical Activity Readiness Questionnaire with one exception: subject will not be excluded if he/she takes a single blood pressure medication that doesn't impact heart rate and blood pressure is controlled on the medication (blood pressure is less than 140/90 mmHg).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jacobs, PhD, Principal Investigator — Oregon Health and Science University; Jessica Castle, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castle JR, Wilson LM, Tyler NS, Espinoza AZ, Mosquera-Lopez CM, Kushner T, Young GM, Pinsonault J, Dodier RH, Hilts WW, Oganessian SM, Branigan DL, Gabo VB, Eom JH, Ramsey K, Youssef JE, Cafazzo JA, Winters-Stone K, Jacobs PG. Assessment of a Decision Support System for Adults with Type 1 Diabetes on Multiple Daily Insulin Injections. Diabetes Technol Ther. 2022 Dec;24(12):892-897. doi: 10.1089/dia.2022.0252. Epub 2022 Sep 5. PMID 35920839

RESULTS

PARTICIPANT FLOW:
Period: Run in Visit Training (2 Hours)
Arm/Group | DailyDose Decision Support
Started | 25
Completed | 25
Not Completed | 0
Period: First at Home Period (~2 Weeks)
Arm/Group | DailyDose Decision Support
Started | 25
Completed | 25
Not Completed | 0
Period: DailyDose Training Visit (2 Hours)
Arm/Group | DailyDose Decision Support
Started | 25
Completed | 25
Not Completed | 0
Period: Second at Home Period (8 Weeks)
Arm/Group | DailyDose Decision Support
Started | 25
Completed | 24
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Study Close-out Visit (30 Minutes)
Arm/Group | DailyDose Decision Support
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DailyDose Decision Support
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Percent of Time With Sensed Glucose Between 70 - 180 mg/dl
Description: Mean change in the percent of time with sensed glucose between 70 - 180 mg/dl based on the Dexcom G6 CGM data between weeks 1-2 and 9-10.
Time Frame: Weeks 1-2 and 9-10
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | DailyDose Decision Support
Number analyzed (Participants) | 24
percentage of time | -3.8 (15.8)

2. Secondary Outcome: Mean Change in Sensed Glucose
Description: Mean change in sensed glucose based on the Dexcom G6 CGM data between weeks 1-2 and 9-10.
Time Frame: Weeks 1-2 and 9-10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DailyDose Decision Support
Number analyzed (Participants) | 24
mg/dL | 11 (28)

3. Secondary Outcome: Mean Change in the Percent of Time With Sensed Glucose <70 mg/dl
Description: Mean change in the percent of time with sensed glucose < 70 mg/dl based on the Dexcom G6 CGM data between weeks 1-2 and 9-10.
Time Frame: Weeks 1-2 and 9-10
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | DailyDose Decision Support
Number analyzed (Participants) | 24
percentage of time | -0.3 (1.0)

4. Secondary Outcome: Mean Change in the Percent of Time With Sensed Glucose <54 mg/dl
Description: Mean change in the percent of time with sensed glucose < 54 mg/dl based on the Dexcom G6 CGM data between weeks 1-2 and 9-10.
Time Frame: Weeks 1-2 and 9-10
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | DailyDose Decision Support
Number analyzed (Participants) | 24
percentage of time | 0.0006 (0.472)

5. Secondary Outcome: Mean Change in the Percent of Time With Sensed Glucose >180 mg/dl
Description: Mean change in the percent of time with sensed glucose >180 mg/dl based on the Dexcom G6 CGM data between weeks 1-2 and 9-10.
Time Frame: Weeks 1-2 and 9-10
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | DailyDose Decision Support
Number analyzed (Participants) | 24
percentage of time | 4.1 (15.9)

6. Secondary Outcome: Mean Change in the Percent of Time With Sensed Glucose >250 mg/dl
Description: Mean change in the percent of time with sensed glucose >250 mg/dl based on the Dexcom G6 CGM data between weeks 1-2 and 9-10.
Time Frame: Weeks 1-2 and 9-10
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | DailyDose Decision Support
Number analyzed (Participants) | 24
percentage of time | 5.4 (12.5)

7. Secondary Outcome: Change in Coefficient of Variation of Sensor Glucose Based on the Dexcom G6 CGM Data.
Description: Change in coefficient of variation of sensor glucose based on the Dexcom G6 CGM data between weeks 1-2 and 9-10.
Time Frame: Weeks 1-2 and 9-10
Measure: Number; unit: percent of CV
Arm/Group | DailyDose Decision Support
Number analyzed (Participants) | 24
percent of CV | -0.3

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: All participants that started a visit are included in the adverse events. All subjects completed all visits except one. That subject only completed two of the three visits.
Arm/Group | DailyDose Decision Support
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DailyDose Decision Support (N=25)
upper respiratory infection (Infections and infestations) | 2 (2)
urinary tract infection (Infections and infestations) | 1 (1)
vaginal infection (Infections and infestations) | 1 (1)
strep throat (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT04428645/Prot_SAP_000.pdf